CLINICAL TRIAL: NCT05144295
Title: Lubiprostone for the Treatment of Functional Constipation in the Under 18 Years Patients: A Randomized, Controlled Trial.
Brief Title: Lubiprostone for Functional Constipation in the Under 18 Years Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Sameh A. Lashen, Associate Professor of Internal Medicine, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0305299
Record Dates: First submitted 2021-11-22; First posted 2021-12-03 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Clinical Efficacy; Treatment Efficacy; Drug Side Effect
Keywords: Lubiprostone; Functional constipation; Adolescent; Children; Spontaneous Bowel Motions; Drug safety
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — Lubiprostone; Capsules; Lactulose; Bisacodyl; picosulfate sodium

STUDY DESIGN:
Intervention Model Description: Patients assigned to lubiprostone will receive a dose based on their weight at the time of enrollment. patients weighing <50 kg and ≥ 50 kg will be given lubiprostone at doses of 8 mg TID and 24 mg BID, respectively.
  Patients and their parents/legal guardians will be instructed to administer the doses at least 5 hours apart with meals and large volume of fluid.
  The control group will receive the conventional therapy (lactulose 1 mL/kg, once or twice daily (maximum 60 mL/day), or Bisacodyl tablet (5 mg/tablet) in a dose of 2 tab/day for < 12 years or 3 tab/day for > 12 years.
  Both arms will receive the treatment for 12 weeks followed by 4 weeks follow-up after the end of treatment (week 16).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Investigational Arm (Experimental): * Patients will receive lubiprostone capsules (Amiprostone 8 and 24 mcg, or Lubicont 8 mcg)
  * Patients weighing <50 kg will be given lubiprostone at doses of 8 mcg/8 hours.
  * Patients weighing ≥ 50 kg will be given lubiprostone at doses of 24 mcg BID.
  * Patients and their parents/legal guardians will be instructed to administer the doses at least 5 hours apart with meals and a large volume of fluid.
  Interventions: Drug: Lubiprostone Pill
- Control Arm (Active Comparator): Subjects will receive the conventional therapy (one or a combination of the following):
  * Lactulose " Lactulose, or Duphalac syrup" at a dose of 1 ml/kg once or twice daily (maximum 60 mL/day),
  * Bisacodyl tablets " Bisacodyl 5 mg/tablet" in a dose of 2 tab/day for < 12 years or 3 tab/day for > 12 years, or
  * Sodium Picosulfate 0.75% drops (Picolax drops) in a daily dose of 2.5-20 mg/day.
  Interventions: Drug: Lactulose Oral Liquid Product; Drug: Bisacodyl 5 MG; Drug: Sodium Picosulfate

INTERVENTIONS:
Drug: Lubiprostone Pill — Oral pills for constipation (Lubiprostone) will be given in a dose range from 24 mcg once daily to 24 mcg twice daily according to the participant weight.
  Other Names: Amiprostone 8 mcg caps; Amiprostone 24 mcg caps; Lubicont 8 mcg caps
  Arms: Investigational Arm
Drug: Lactulose Oral Liquid Product — Lactulose " Lactulose, or Duphalac syrup" at a dose of 1 ml/kg once or twice daily (maximum 60 mL/day)
  Other Names: Lactulose OR Duphalac
  Arms: Control Arm
Drug: Bisacodyl 5 MG — Bisacodyl tablet (5 mg/tablet) in a dose of 2 tab/day for < 12 years or 3 tab/day for > 12 years
  Other Names: Bisacodyl 5 mg tablets
  Arms: Control Arm
Drug: Sodium Picosulfate — Sodium Picosulfate 0.75% drops in a daily dose of 2.5-20 mg/day
  Other Names: Bisadyl 0.75% drops
  Arms: Control Arm

SUMMARY:
The investigators will enroll subjects 8 - < 18 years of age, fulfilling Rome IV criteria for functional constipation.

Participants will be randomly assigned to either Lubiprostone treatment (study group), or the control group (will receive either lactulose or Bisacodyl tablets).

safety and efficacy will be assessed.

DETAILED DESCRIPTION:
The investigators will enroll 274 subjects who will be randomly divided equally into interventional and control groups.

Participants and their parents/legal guardians will be instructed to administer the doses at least 5 hours apart with meals and a large volume of fluid.

The control group will receive lactulose 1 mL/kg, once or twice daily (maximum 60 mL/day or Bisacodyl tablet (5 mg/tablet) in a dose of 2 tab/day for < 12 years or 3 tab/day for > 12 years.

Both arms will receive the treatment for 12 weeks followed by 4 weeks follow-up after the end of treatment (week 16).

Participants (and their guardians) will be instructed to regularly document the number of spontaneous bowel motions/week and to define their Bristol chart category for every bowel motion. In addition, the participants will be encouraged to contact the trial team if any adverse events appeared. This is in addition to regular visits at 0, 2, 8, 12 weeks for assessment of safety (efficacy will be assessed at weeks 8, 12, and 16).

ELIGIBILITY:
Inclusion Criteria:

* Patients 8 - < 18 years of age who have a confirmed diagnosis of Pediatric functional constipation according to the Rome IV criteria, who give written informed consent personally or from their legal guardians.
* Discontinuation of any medication affecting gastrointestinal (GI) motility at least 2 weeks before starting the treatment allocation.
* Patient's daily diary that indicates an average of < 3 weekly spontaneous bowel movements (SBMs), with ≥ 25% of SBMs involving at least some straining and/or a 5-point modified Bristol Stool Form Scale type 1 or 2.
* Patients who completed the study protocol.

Exclusion Criteria:

1. If the patient's constipation is attributed to any of the following: physical, mental, or cognitive illness, inflammatory bowel disease, medication, anatomical, neurological, endocrine, or metabolic factors.
2. If the patient is a candidate for or underwent abdominal surgery, or has any condition other than constipation that could affect gastrointestinal motility or defecation.
3. Patients suffering from Hirschsprung's disease.
4. Patients experiencing any alarming signs e.g. unexplained significant weight loss.
5. Untreated fecal impaction at the time of enrollment.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 274 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-08-25 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Primary outcome | At study week 16.
  Spontaneous bowel motions (SBM) ≥ 1 SBM/week increase in the frequency compared with baseline, and ≥ 3 SBMs/week for at least 8 weeks, including the last 4 study weeks and the 4 weeks of follow-up.

SECONDARY OUTCOMES:
Early spontaneous bowel motions | First 48 hours after first drug dose.
  Number of participants who experienced first SBM within 48 hours after dose initiation.
First dose response time | 1st week of treatment
  The time between first dose of treatment and the first SBM.
Number of Spontaneous Bowel Motions/Week. | At study week Week 8, 12.
  Number of Spontaneous Bowel Motions/Week.
Responders rate | At study week Week 8, 12, 16.
  Responders rate at week 8, 12, 16.

CONTACTS AND LOCATIONS:
Overall Officials: Sameh A. Lashen, MD (Ph.D.), Principal Investigator — Faculty of Medicine, Alexandria University - Alexandria
Locations (2):
- Egypt (2):
  - Alexandria Main University Hospital, Alexandria
  - Faculty of Medicine, Alexandria

IPD SHARING:
Plan to Share IPD: No
patient personal and identification data will not be available for sharing